CLINICAL TRIAL: NCT03808584
Title: Impact of Core Muscle Training on Incisional Hernia and Pain After Abdominal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018-00958
Record Dates: First submitted 2019-01-15; First posted 2019-01-17 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Hernia Incisional; Exercise
Keywords: Core muscle exercise; rehabilitation; Incisional hernia
MeSH Terms: conditions — Incisional Hernia; Motor Activity | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The patients in the control group will receive standard physiotherapy and will be instructed to limit core muscle activity and weight bearing according to their pain symptomatology. Standard physiotherapy for all hospitalised patients includes early mobilization and exercises to prevent thrombosis and pulmonary complications (atelectasis, pneumonia, diaphragmatic deconditioning), balance training and endurance and exercise training
- Intervention group (Experimental): The patients in the intervention group will be given exercises to perform postoperatively.They will be instructed by a physiotherapist in how to perform the four specific exercises targeting core muscles. The patient will perform these exercises daily during hospitalization under the supervision of the physiotherapist and then at home for two months after the operation. The intensity of the exercises will be adjusted daily to the physical capabilities of the patient. They will also benefit from standard physiotherapy as described above.
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Physiotherapy — 4 specific core muscle exercises, targeting abdominal muscles, to be performed daily from postoperative day one to 2 months postsurgery.
  Arms: Intervention group

SUMMARY:
The current practice to avoid incisional hernia, one of the most frequent complications following abdominal surgery, is to minimize core muscle activity in the postoperative phase. However, there is no evidence to support the association of core muscle activity and increased incidence of incisional hernia. On the contrary, it is likely that reduced physical activity could lead to physical deconditioning, chronic postsurgical pain (CPSP), and sarcopenia. The investigators will conduct a prospective multicentric randomized clinical trial to compare standard of care to core muscle exercises targeting the abdominal muscles immediately postsurgery. The principle hypothesis is that neither specific exercises of core muscles before and after surgery nor physical restriction alter the incidence of incisional hernias. Secondly the impact of postoperative rehabilitation on CPSP and sarcopenia will be assessed.

DETAILED DESCRIPTION:
The current practice to avoid incisional hernia, one of the most frequent complications following abdominal surgery, is to minimize core muscle activity in the postoperative phase. Therefore the patients are instructed not to bear or lift weights and to limit physical activities in the first 8-12 weeks after surgery. However, there is no evidence to support the association of core muscle activity and increased incidence of incisional hernia. On the contrary, it is likely that reduced physical activity and deconditioning of the core muscles is associated with muscle catabolism, which may lead to physical deconditioning, chronic postsurgical pain (CPSP), and sarcopenia. CPSP is primarily a major burden in terms of reduced quality of life and resource utilization whereas sarcopenia in addition is increasingly recognized as an important independent risk factor for numerous adverse clinical outcomes and mortality.

The investigators will conduct a prospective multicentric randomized clinical trial to compare standard of care to core muscle exercises targeting the abdominal muscles immediately postsurgery. The principle hypothesis is that neither specific exercises of core muscles before and after surgery nor physical restriction alter the incidence of incisional hernias. Secondly the impact of postoperative rehabilitation on CPSP and sarcopenia will be assessed. The patients will be divided into two study arms, one receiving standard of care and the other receiving the intervention. The intervention consists of four specific core muscle exercises to perform daily during the first two months after surgery. Follow-up will be at two, twelve and twenty-four months with clinical examination and ultrasound to detect incisional hernias, assessment chronic postsurgical pain and its treatment and evaluation of muscle mass on CT scans.

ELIGIBILITY:
Inclusion Criteria:

1. At the University Hospital of Bern, Kantonsspital Solothurn and Olten and BundeswehrZentralkrankenhaus Koblenz:

   * Informed Consent as documented by signature (Appendix Informed Consent Form)
   * Age > 18 years
   * Capable of judgment
   * Undergoing elective or emergency abdominal surgery
   * Laparoscopic or open surgery, midline or transverse incision
2. At the University Hospital of Lausanne:

   * Informed Consent as documented by signature (Appendix Informed Consent Form)
   * Age > 18 years
   * Capable of judgment
   * Undergoing elective open abdominal surgery
   * Midline or transverse incision

Exclusion criteria (in all four participating centres):

* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders (chronic depression, under antidepressants or neuroleptics), dementia, etc. of the participant
* Enrolment of the investigator, his/her family members, employees and other dependent persons
* Neuromuscular diseases (such as myasthenia gravis or wheelchair-bound patient)
* Preexisting chronic pain disorder, patients under chronic opioid therapy (WHO II and III) or pain modulating drugs (antidepressive medication or antiepileptic medication)
* End-stage disease
* Patients with preexisting abdominal wall mesh, with the exception of inguinal mesh (after inguinal hernia repair)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 588 (Estimated)
Dates: Start 2019-05-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of incisional hernia 24 months postsurgery | 24 months postsurgery
  Incidence of incisional hernia diagnosed by ultrasound and clinical examination

SECONDARY OUTCOMES:
Incidence of Chronic postsurgical pain | 2 months, 12 months, 24 months after surgery
  Abdominal pain assessment by Visual Analog Scale (VAS). VAS score ranges from 0 (no pain) to 10 (worst possible pain). The mean VAS in the last 24 hours will be documented.
Exercise | 2 days after surgery, at discharge, 2 months after surgery
  Exercise type and number of repetitions
Length of hospital stay | End of hospital stay, expected to be up to 4 weeks
  Length of hospital stay
Readmission rate | 2 months, 12 months, 24 months after surgery
  Hospital readmission
Re-operation rate | 2 months, 12 months, 24 months after surgery
  Re-operation
Incidence of Sarcopenia | 2 months and 24 months after surgery
  Muscle mass as assessed by comparing preoperative and postoperative CT scans in subgroup of patients who underwent these examinations for other medical reasons

CONTACTS AND LOCATIONS:
Overall Officials: Guido Beldi, MD, Study Director — Department for visceral surgery, University Hospital Bern, Inselspital, Switzerland
Locations (5):
- BundeswehrZentralkrankenhaus, Koblenz, Germany
- Switzerland (4):
  - Kantonsspital Olten, Olten, Canton of Solothurn
  - University Hospital of Bern, Inselspital, Bern
  - CHUV, University Hospital of Lausanne, Lausanne
  - Bürgerspital Solothurn, Solothurn

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pommergaard HC, Burcharth J, Danielsen A, Angenete E, Haglind E, Rosenberg J. No consensus on restrictions on physical activity to prevent incisional hernias after surgery. Hernia. 2014 Aug;18(4):495-500. doi: 10.1007/s10029-013-1113-8. Epub 2013 May 28. PMID 23712287
- [Background] Katsura M, Kuriyama A, Takeshima T, Fukuhara S, Furukawa TA. Preoperative inspiratory muscle training for postoperative pulmonary complications in adults undergoing cardiac and major abdominal surgery. Cochrane Database Syst Rev. 2015 Oct 5;2015(10):CD010356. doi: 10.1002/14651858.CD010356.pub2. PMID 26436600
- [Background] Bruce J, Krukowski ZH. Quality of life and chronic pain four years after gastrointestinal surgery. Dis Colon Rectum. 2006 Sep;49(9):1362-70. doi: 10.1007/s10350-006-0575-5. PMID 16741597
- [Background] Otsuji H, Yokoyama Y, Ebata T, Igami T, Sugawara G, Mizuno T, Yamaguchi J, Nagino M. Surgery-Related Muscle Loss and Its Association with Postoperative Complications After Major Hepatectomy with Extrahepatic Bile Duct Resection. World J Surg. 2017 Feb;41(2):498-507. doi: 10.1007/s00268-016-3732-6. PMID 27718001
- [Result] Itatsu K, Yokoyama Y, Sugawara G, Kubota H, Tojima Y, Kurumiya Y, Kono H, Yamamoto H, Ando M, Nagino M. Incidence of and risk factors for incisional hernia after abdominal surgery. Br J Surg. 2014 Oct;101(11):1439-47. doi: 10.1002/bjs.9600. Epub 2014 Aug 14. PMID 25123379